CLINICAL TRIAL: NCT05584566
Title: Ridge Augmentation Treatment Using OSSIX® BREEZE vs Jason® Membrane in Simultaneous Implantations. A Prospective, Randomized Controlled Trial.
Brief Title: Ridge Augmentation Treatment Using OSSIX® BREEZE vs Jason®
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Datum Dental LTD (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: DD-OG-01
Record Dates: First submitted 2022-10-11; First posted 2022-10-18 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Ridge Augmentation

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OSSIX Breeze (Experimental)
  Interventions: Device: OSSIX Breeze
- Jason membrane (Active Comparator)
  Interventions: Device: Jason membrane

INTERVENTIONS:
Device: OSSIX Breeze — barrier membrane
  Arms: OSSIX Breeze
Device: Jason membrane — barrier membrane
  Arms: Jason membrane

SUMMARY:
This is a prospective randomized controlled parallel trial. The aim of this study is to evaluate bone formation and soft tissue healing after 4 and 8 months in patients with ridge deficiencies in simultaneous implantation approach. The trial will compare a (sugar cross linked) - SCL pericardium membrane OSSIX® Breeze vs native pericardium membrane (Jason®).

ELIGIBILITY:
Inclusion Criteria:

1. Males and females, age 18 and above.
2. General good health (ASA 1 and ASA 2).
3. Adults with buccal bone defect, who are in need of implant placement, and going through a guided bone regeneration treatment.
4. Patient needs 1-3 implants.
5. Good oral hygiene (full mouth plaque index <25%).
6. Adequate control of inflammation (full mouth bleeding on probing <25%).
7. Patient is willing to sign an informed consent and participate in the clinical study.

10 8. Patient is able to understand and comply with the study related procedures, such as exercising good oral hygiene and attending all follow-up examinations.

Exclusion Criteria:

1. Physical status ASA III or ASA IV.
2. General contraindications for dental and/or surgical treatments.
3. Inflammatory and autoimmune disease of the oral cavity.
4. Patients with known collagen hypersensitivity.
5. Patients with sensitivity to porcine-derived materials.
6. Patients suffering from autoimmune diseases and connective tissue diseases, such as: systemic lupus erythematosus, dermatomyositis, etc.
7. Acute infection in the oral cavity or acute inflammation at the implantation site.
8. General diseases, where measures of stomatology, maxillo-facial surgery, implantology, periodontology, endodontology or other measures of oral surgery are contraindicated.
9. Disease of oral mucosa.
10. Uncontrolled periodontal disease
11. Concurrent or previous radiotherapy of head area.
12. Concurrent or previous immunosuppressant, bisphosphonate, or high-dose corticosteroid therapy.
13. Smoking (over 10 cigarettes a day).
14. Pregnant or lactating women.
15. Women of childbearing potential, who are not using a highly effective method of birth control.
16. Participation in another investigational device, drug, or biologics study within the last 24 weeks prior to study entry.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2026-06-01 (Estimated); Study Completion 2026-07-01 (Estimated)

PRIMARY OUTCOMES:
increase in bone gain | 4 months
  increase in bone gain (vertical and horizontal) in mm, 4 months after the implant placement in the augmented site. the measurment will be done according to radiographic images

CONTACTS AND LOCATIONS:
Locations (3):
- Israel (2):
  - Hadassah Medical Center, Jerusalem
  - Rabin Medical Center, Petah Tikva
- University of Birmingham, Birmingham, United Kingdom